CLINICAL TRIAL: NCT06254287
Title: Efficacy and Safety of Avatrombopag vs. Avatrombopag Combined With rhTPO in the Treatment of Patients With Severe Aplastic Anemia
Brief Title: Efficacy and Safety of Avatrombopag vs. Avatrombopag Combined With rhTPO in the Treatment of SAA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Fosun Pharmaceutical Distribution Jiangsu co., Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKX-AA-001
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-10

CONDITIONS: Anemia, Aplastic
Keywords: Aplastic anemia，Avatrombopag，rhTPO，Efficacy，Safety
MeSH Terms: conditions — Anemia, Aplastic | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Avatrombopag group (Experimental): The Avatrombopag group was given Avatrombopag: 40 mg/ time, once a day, orally, for 3 months
  Interventions: Drug: Avatrombopag
- Avatrombopag +rhTPO group (Other): Avatrombopag: 40 mg/ time, once a day, orally; rhTPO: 15000U/ time, once a day, subcutaneous injection; Both were 3 months.
  Interventions: Drug: Avatrombopag +rhTPO

INTERVENTIONS:
Drug: Avatrombopag — Avatrombopag was given 40 mg/ time, once a day, orally, for 3 months.
  Arms: Avatrombopag group
Drug: Avatrombopag +rhTPO — Avatrombopag: 40 mg/ time, once a day, orally; rhTPO: 15000U/ time, once a day, subcutaneous injection; Both were 3 months.
  Arms: Avatrombopag +rhTPO group

SUMMARY:
Title: Efficacy and safety of Avatrombopag VS Avatrombopag combined with rhTPO in patients with severe aplastic anemia: a single-center, controlled study Observation group: Patients with severe aplastic anemia who did not respond to initial treatment (unconditional HSCT or ATG) or other treatments (except HSCT) Objective: To evaluate the efficacy and safety of Avatrombopag and rhTPO in the treatment of patients with severe aplastic anemia, to provide more treatment options for patients with severe aplastic anemia who are unable to undergo transplantation /ATG or have failed previous treatment, and to provide evidence-based evidence for the use of Avatrombopag or combined with rhTPO to promote hematopoietic recovery Experimental design: Single center, controlled study Total number of cases: 30 cases/group, 2 groups

Case selection criteria:

Inclusion criteria:

1. Age: > 18 years old, gender is not limited;
2. Patients clinically diagnosed with severe aplastic anemia (diagnostic criteria: ① myelocyte hyperplasia < 25% of normal; If ≥ 25% of normal but < 50%, the remaining hematopoietic cells should be < 30%. ② Blood routine must have two of the following three items: ANC < 0.5×109 /L; The absolute value of reticulocyte was < 20×109 /L; PLT < 20×109 /L). ③ If ANC < 0.2×109 /L, the diagnosis is very severe aplastic anemia), including patients who are newly diagnosed or have failed other treatments;
3. Patients currently undergoing hematopoietic stem cell transplantation or ATG without conditions;
4. Eastern Cancer Collaboration Group (ECOG) score 0-2;
5. Informed consent must be signed before participating in the study.

Exclusion criteria:

One of the following circumstances is not eligible for inclusion:

1. Patients with severe bleeding and/or infection that cannot be controlled after standard treatment;
2. Diagnosis of congenital hematopoietic failure (such as Fanconi anemia, congenital dyskeratosis, etc.);
3. Other causes of pancytopenia and bone marrow hypoproliferative diseases (such as hemolytic PNH, hypoproliferative MDS/AML, autoantibody-mediated pancytopenia, etc.);
4. All laboratory or clinically confirmed HIV infection, hepatitis C infection, chronic hepatitis B infection, or evidence of active hepatitis during screening;
5. Cytogenetic evidence of bone marrow abnormalities in clonal blood diseases;
6. History of thromboembolism or current use of anticoagulants within the past 6 months;
7. Accompanied by any one or more malignant diseases;
8. Treatment with another investigational agent within 30 days prior to the first dose of Avatrombopag;
9. Patients who cannot understand or are unwilling to sign an informed consent form (ICF);
10. Pregnant or lactating women;
11. The female patient or the female spouse of the male patient is unable to take effective contraceptive measures;
12. The Investigator considers that there are any other circumstances that may cause the subject to be unable to complete the study or that pose a significant risk to the subject.

Exit criteria:

1. The subject or his legal guardian voluntarily requests withdrawal;
2. Violation of inclusion/exclusion criteria;
3. Poor medication compliance;
4. The subject's condition requires treatment with drugs prohibited by the study;
5. Adverse events occur that cause subjects to be unable to continue the study;
6. Other unexplained severe comorbidities;
7. Pregnancy occurs during treatment;
8. Subjects deemed unsuitable for further study by the investigator.

Test termination:

1. For safety reasons, the study sponsor proposes to stop the study;
2. The Ethics committee decides to stop the study;
3. The lead researcher decides to stop the study. Investigational drug: Avatrombopag: tablet, specification: 20 mg/ tablet. rhTPO: 15000 units /1 ml. Treatment plan: This clinical trial is planned to carry out a 3-month drug study.

A: The Avatrombopag group was given Avatrombopag: 40 mg/ time, once a day, orally, for 3 months.

B: Avatrombopag +rhTPO group, Avatrombopag: 40 mg/ time, once a day, orally; rhTPO: 15000U/ time, once a day, subcutaneous injection; Both were 3 months.

Efficacy index:

Main therapeutic indicators:

Overall response rate at 3 months (OR);

Secondary efficacy measures:

Complete response rate at 3 months (CR); The time of the first occurrence of PR and CR within 3 months of medication; The proportion of subjects who were off platelet transfusion at 3 months; Hemorrhage score records of patients within 3 months of medication; Health-related quality of life score (SF-36 scale).

Efficacy criteria:

Complete response (CR) : HGB > 100 g/L; ANC > 1.5 × 109 /L; PLT > 100×109/L; Partial response (PR) : disengagement from component blood transfusion and no longer meeting the diagnostic criteria for SAA; Invalid (NR) : SAA diagnostic criteria are still met.

DETAILED DESCRIPTION:
Title: Efficacy and safety of Avatrombopag VS Avatrombopag combined with rhTPO in patients with severe aplastic anemia: a single-center, controlled study Version number: V3.0 Observation group: Patients with severe aplastic anemia who did not respond to initial treatment (unconditional HSCT or ATG) or other treatments (except HSCT) Objective: To evaluate the efficacy and safety of Avatrombopag and rhTPO in the treatment of patients with severe aplastic anemia, to provide more treatment options for patients with severe aplastic anemia who are unable to undergo transplantation /ATG or have failed previous treatment, and to provide evidence-based evidence for the use of Avatrombopag or combined with rhTPO to promote hematopoietic recovery Experimental design: Single center, controlled study Total number of cases: 30 cases/group, 2 groups

Case selection criteria:

Inclusion criteria:

1. Age: > 18 years old, gender is not limited;
2. Patients clinically diagnosed with severe aplastic anemia (diagnostic criteria: ① myelocyte hyperplasia < 25% of normal; If ≥ 25% of normal but < 50%, the remaining hematopoietic cells should be < 30%. ② Blood routine must have two of the following three items: ANC < 0.5×109 /L; The absolute value of reticulocyte was < 20×109 /L; PLT < 20×109 /L). ③ If ANC < 0.2×109 /L, the diagnosis is very severe aplastic anemia), including patients who are newly diagnosed or have failed other treatments;
3. Patients currently undergoing hematopoietic stem cell transplantation or ATG without conditions;
4. Eastern Cancer Collaboration Group (ECOG) score 0-2;
5. Informed consent must be signed before participating in the study.

Exclusion criteria:

One of the following circumstances is not eligible for inclusion:

1. Patients with severe bleeding and/or infection that cannot be controlled after standard treatment;
2. Diagnosis of congenital hematopoietic failure (such as Fanconi anemia, congenital dyskeratosis, etc.);
3. Other causes of pancytopenia and bone marrow hypoproliferative diseases (such as hemolytic PNH, hypoproliferative MDS/AML, autoantibody-mediated pancytopenia, etc.);
4. All laboratory or clinically confirmed HIV infection, hepatitis C infection, chronic hepatitis B infection, or evidence of active hepatitis during screening;
5. Cytogenetic evidence of bone marrow abnormalities in clonal blood diseases;
6. History of thromboembolism or current use of anticoagulants within the past 6 months;
7. Accompanied by any one or more malignant diseases;
8. Treatment with another investigational agent within 30 days prior to the first dose of Avatrombopag;
9. Patients who cannot understand or are unwilling to sign an informed consent form (ICF);
10. Pregnant or lactating women;
11. The female patient or the female spouse of the male patient is unable to take effective contraceptive measures;
12. The Investigator considers that there are any other circumstances that may cause the subject to be unable to complete the study or that pose a significant risk to the subject.

Exit criteria:

1. The subject or his legal guardian voluntarily requests withdrawal;
2. Violation of inclusion/exclusion criteria;
3. Poor medication compliance;
4. The subject's condition requires treatment with drugs prohibited by the study;
5. Adverse events occur that cause subjects to be unable to continue the study;
6. Other unexplained severe comorbidities;
7. Pregnancy occurs during treatment;
8. Subjects deemed unsuitable for further study by the investigator.

Test termination:

1. For safety reasons, the study sponsor proposes to stop the study; 2. The Ethics committee decides to stop the study; 3. The lead researcher decides to stop the study. Investigational drug: Avatrombopag: tablet, specification: 20 mg/ tablet. rhTPO: 15000 units /1 ml. Treatment plan: This clinical trial is planned to carry out a 3-month drug study.

A: The Avatrombopag group was given Avatrombopag: 40 mg/ time, once a day, orally, for 3 months.

B: Avatrombopag +rhTPO group, Avatrombopag: 40 mg/ time, once a day, orally; rhTPO: 15000U/ time, once a day, subcutaneous injection; Both were 3 months.

Dose adjustment:

A: In the Avatrombopag group, if PLT≥200×109 /L lasted for 2 weeks or ≥100×109 /L lasted for 1 month, the dosage of Avatrombopag was reduced to 20 mg/d; If PLT remained ≥200×109 /L for 2 weeks or ≥100×109 /L for 1 month, the dosage of Avatrombopag was reduced to 20 mg once every other day. If the PLT is still ≥200×109/L for 2 weeks or ≥100×109 /L for 1 month, the drug should be stopped. If PLT rose rapidly and was ≥400×109 /L, the drug should be stopped and observed until PLT < 100×109 /L, and then continued with 20 mg/d.

B: Avatrombopag group +rhTPO: dosage adjustment of Avatrombopag as above; If PLT rises to ≥100×109/L for 2 weeks, rhTPO will be reduced to 15000u every other day. If PLT is still ≥100×109/L for 2 weeks, rhTPO will be reduced to 15000u every 3 days. If the PLT is still ≥100×109/L for 2 weeks, stop.

Efficacy index:

Main therapeutic indicators:

Overall response rate at 3 months (OR);

Secondary efficacy measures:

Complete response rate at 3 months (CR); The time of the first occurrence of PR and CR within 3 months of medication; The proportion of subjects who were off platelet transfusion at 3 months; Hemorrhage score records of patients within 3 months of medication; Health-related quality of life score (SF-36 scale).

Efficacy criteria:

Complete response (CR) : HGB > 100 g/L; ANC > 1.5 × 109 /L; PLT > 100×109/L; Partial response (PR) : disengagement from component blood transfusion and no longer meeting the diagnostic criteria for SAA; Invalid (NR) : SAA diagnostic criteria are still met.

Safety indicators:

1. Incidence of clonal evolution at 1 and 2 years after treatment, including clonal evolution to PNH, and evolution to AML or MDS;
2. Adverse events (evaluated according to the Evaluation Criteria for Common Adverse Events (CTCAE) version 5.0), laboratory tests, vital signs, electrocardiogram records and physical examination, etc., were evaluated for the safety of the tested drug.

Study process: Screening period (-7-0 days)

1. Obtain informed consent;
2. Collect demographic information and basic data of subjects;
3. Record the medical history and current treatment, and combine drugs;
4. Vital signs, physical examination;
5. Blood test: blood routine and blood biochemistry (including liver and kidney function);
6. Bone marrow puncture and biopsy;
7. Pregnancy test (for women of childbearing age);
8. Review the entry criteria. Visit 1 (+1 day) After baseline screening, patients meeting the inclusion criteria were given medication at baseline according to group A and Group B, respectively.

1. Blood test: blood routine and blood biochemistry (including liver and kidney function); 2. Vital signs and physical examination; 3. Record drug combinations, including blood transfusion; 4. Bleeding score was recorded; 5. Health-related quality of life score; 6. Record adverse events after medication. Visit 2 (+2 weeks)

1. Blood test: blood routine and blood biochemistry (including liver and kidney function);
2. Vital signs and physical examination;
3. Record drug combinations, including blood transfusion;
4. Bleeding score was recorded;
5. Health-related quality of life score;
6. Record adverse events after medication. Visit 3 (+4 weeks)

1. Blood test: blood routine and blood biochemistry (including liver and kidney function); 2. Vital signs and physical examination; 3. Record drug combinations, including blood transfusion; 4. Bleeding score was recorded; 5. Health-related quality of life score; 6. Record adverse events after medication. Visit 4 (+6 weeks)

1. Blood test: blood routine and blood biochemistry (including liver and kidney function);
2. Vital signs and physical examination;
3. Record drug combinations, including blood transfusion;
4. Bleeding score was recorded;
5. Health-related quality of life score;
6. Record adverse events after medication. Visit 5 (+8 weeks)

1. Blood test: blood routine and blood biochemistry (including liver and kidney function); 2. Vital signs and physical examination; 3. Record drug combinations, including blood transfusion; 4. Bleeding score was recorded; 5. Health-related quality of life score; 6. Record adverse events after medication. Visit 6 (+10 weeks)

1. Blood test: blood routine and blood biochemistry (including liver and kidney function);
2. Vital signs and physical examination;
3. Record drug combinations, including blood transfusion;
4. Bleeding score was recorded;
5. Health-related quality of life score;
6. Record adverse events after medication. Visit 7 (+12 weeks /3 months)

1. Blood test: blood routine and blood biochemistry (including liver and kidney function); 2. Vital signs and physical examination; 3. Record drug combinations, including blood transfusion; 4. Bleeding score was recorded; 5. Health-related quality of life score; 6. Record adverse events after medication; 7. Pregnancy test (for women of childbearing age); 8. Genetic examination to analyze chromosome mutations; 9. Bone marrow puncture and biopsy. Long-term follow-up is recommended for patients with conditions. Adverse events were closely observed during the study, and the combination of drugs was recorded in detail.

Drug combination:

1. Platelet transfusion is allowed according to clinical bleeding conditions: patients with PLT < 20×109/L, patients with stable PLT < 10×109/L, or patients with severe bleeding can be supported by platelet suspension collected by infusion machine;
2. Erythrocyte transfusion can be considered when hemoglobin < 60 g/L;
3. For those who need Shengbai injection after clinical evaluation, G-CSF should be given 150-600ug/d;
4. For drugs that have been used before the test, try to maintain the original dose during the test;
5. From the signing of informed consent to the end of the trial, all subjects were examined for adverse events and accompanying medications at each visit;
6. All drug combinations should be recorded in the column of drug combinations in the Case observation form (CRF) and explained.

Statistical analysis:

Statistical analysis method:

SPSS 26.0 software was used for statistical analysis. The measurement data were described statistically by means of ± standard deviation. The changes before and after treatment were compared with the baseline values using paired T-test. Changes before and after treatment were compared using analysis of variance (ANOVA) or Wilcoxon rank sum test. Counting data were statistically described by frequency (component ratio). All statistical tests were carried out using bilateral tests, and the statistical quantity and exact probability P-value were given. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 18 years old, gender is not limited;
2. Patients clinically diagnosed with severe aplastic anemia (diagnostic criteria: ① myelocyte hyperplasia < 25% of normal; If ≥ 25% of normal but < 50%, the remaining hematopoietic cells should be < 30%. ② Blood routine must have two of the following three items: ANC < 0.5×109 /L; The absolute value of reticulocyte was < 20×109 /L; PLT < 20×109 /L). ③ If ANC < 0.2×109 /L, the diagnosis is very severe aplastic anemia), including patients who are newly diagnosed or have failed other treatments;
3. Patients currently undergoing hematopoietic stem cell transplantation or ATG without conditions;
4. Eastern Cancer Collaboration Group (ECOG) score 0-2;
5. Informed consent must be signed before participating in the study.

Exclusion Criteria:

One of the following circumstances is not eligible for inclusion:

1. Patients with severe bleeding and/or infection that cannot be controlled after standard treatment;
2. Diagnosis of congenital hematopoietic failure (such as Fanconi anemia, congenital dyskeratosis, etc.);
3. Other causes of pancytopenia and bone marrow hypoproliferative diseases (such as hemolytic PNH, hypoproliferative MDS/AML, autoantibody-mediated pancytopenia, etc.);
4. All laboratory or clinically confirmed HIV infection, hepatitis C infection, chronic hepatitis B infection, or evidence of active hepatitis during screening;
5. Cytogenetic evidence of bone marrow abnormalities in clonal blood diseases;
6. History of thromboembolism or current use of anticoagulants within the past 6 months;
7. Accompanied by any one or more malignant diseases;
8. Treatment with another investigational agent within 30 days prior to the first dose of Avatrombopag;
9. Patients who cannot understand or are unwilling to sign an informed consent form (ICF);
10. Pregnant or lactating women;
11. The female patient or the female spouse of the male patient is unable to take effective contraceptive measures;
12. The Investigator considers that there are any other circumstances that may cause the subject to be unable to complete the study or that pose a significant risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
OR | 3 months
  Overall response rate at 3 months

SECONDARY OUTCOMES:
CR | 3 months
  Complete response rate at 3 months
The time of the first occurrence of PR and CR within 3 months of medication | within 3 months of medication
  The time of the first occurrence of PR and CR within 3 months of medication
The proportion of subjects who were off platelet transfusion at 3 months | 3 months
  The proportion of subjects who were off platelet transfusion at 3 months
Hemorrhage score records | within 3 months of medication
  Hemorrhage score records of patients within 3 months of medication
SF-36 scale | 12 months
  Health-related quality of life score (SF-36 scale)

IPD SHARING:
Plan to Share IPD: No